CLINICAL TRIAL: NCT07361224
Title: CLS-015-TAMSC-LBCL-PR An Exploratory, Investigator Initiated Study to Assess the Safety of Combination of CLS-015 (DFF) With Anti-CD-19 CAR-T Cells in Patients With Stable/ Progressive Large B Cell Lymphoma at Lymphodepletion.
Brief Title: Investigator Initiated Study to Assess the Safety of Combination of CLS-015 With Anti-CD-19 CAR-T Cells in Patients With Stable/Progressive Large B Cell Lymphoma at Lymphodepletion.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0126-25
Record Dates: First submitted 2026-01-04; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Large B-Cell Lymphoma (LBCL)
Keywords: Large B-Cell lymphoma
MeSH Terms: interventions — dornase alfa

STUDY DESIGN:
Intervention Model Description: CLS-015 (Dornase Alpha; DFF) is a recombinant human DNase I (rhDNase I), designed to degrade NETs both at the tumor tissue and in systemic blood circulation. CLS-015 increases performance of anti-CD19 CAR-T therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLS-015 infusions after CAR-T infusion (Experimental): CLS-015 infusions will be done on Days 0,3,6,10 and 15 after CAR-T infusion
  Interventions: Drug: rhDNase I

INTERVENTIONS:
Drug: rhDNase I — CLS-015 IV infusions after CAR-T infusion done on Days 0,3,6,10 and 15 after CAR-T infusion

SUMMARY:
This is a Phase 1, single-center, open-label study to evaluate the safety of CLS-015 in combination with anti-CD19 CAR-T therapy in patients with large B-cell lymphoma. The goal is to improve clinical response by reversing the negative effects of NETs on immune function and CAR-T cells.

DETAILED DESCRIPTION:
Disease progression in large B-cell lymphoma is a major obstacle to successful CAR-T therapy, with approximately 40% of patients experiencing disease progression within 3 months of CAR-T infusion and 60% of patients experiencing disease progression within the first year.

While patients with large B-cell lymphoma in partial response or complete response during lymphodepletion have a progression-free survival (PFS) of 60-80% at 1 year, patients with stable disease (SD) or progressive disease (PD) in the lymphodepletion phase have a poor PFS of 20-30%.

Patients with SD/PD in the lymphoid depletion phase, particularly those with low CAR-T concentrations on day +7, are at very high risk of early disease progression after CAR-T infusion, and there is an urgent and unmet medical need to improve their outcomes.

Preclinical studies have shown that CLS-015 enhances the performance of CAR T-cell therapy against CD19-expressing malignancies through various mechanisms, including enhancing CAR T-cell activity, preventing T-cell exhaustion, reducing cytokine release syndrome (CRS), and enhancing CAR-T cell penetration into areas with lymphoma cells by enzymatically degrading NETs in tumor tissue and the bloodstream.

All patients enrolled in the study with large B-cell lymphoma in SD/PD during lymphodepletion will receive CLS-015 on days 0, 3, 6, 10, and 15 after CAR-T cell infusion, as an intravenous infusion.

Patient will be followed for blood test, incidence and severity of cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity (ICANS), immune effector cell-associated HLH-like syndrome (IEC-HS), and cytopenias.

Follow up in the study will be done daily for 15 days post CAR-T infusion, then twice weekly for 15 more days. More checkups will be done at 2-, 6-, 9- and 12-months post CAR-T infusion.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age inclusive, at the time of signing the informed consent.
* Large B-Cell lymphoma treated with CAR-T targeting CD19 (tisagenlecleucel, axicabtagene ciloleucel, or lisocabtagene maraleucel)
* Stable Disease or Progressive Disease confirmed by PET-CT on the day of lymphodepletion
* Capable of giving signed informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

* Hypersensitivity to CLS-015
* Evidence of any clinically significant condition, disorder, condition, or disease that, in the opinion of the Investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Active infection requiring antibiotics
* Females only: Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CLS-015 in combination with anti CD19 CAR T therapy in subjects with stable/progressive Large B-Cell lymphoma at lymphodepletion when CLS-015 is given in adjuvant setting. | Through study completion, an average of 2 years.
  Safety and tolerability of CLS-015 based on adverse events evaluation and recording will be evaluated from screening to the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Ram, Prof., Principal Investigator — Sourasky Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
The plan for sharing individual participant data has not yet been determined at this time

REFERENCES:
- [Background] Nie M, Yang L, Bi X, Wang Y, Sun P, Yang H, Liu P, Li Z, Xia Y, Jiang W. Neutrophil Extracellular Traps Induced by IL8 Promote Diffuse Large B-cell Lymphoma Progression via the TLR9 Signaling. Clin Cancer Res. 2019 Mar 15;25(6):1867-1879. doi: 10.1158/1078-0432.CCR-18-1226. Epub 2018 Nov 16. PMID 30446590
- [Background] Borghaei H, Gettinger S, Vokes EE, Chow LQM, Burgio MA, de Castro Carpeno J, Pluzanski A, Arrieta O, Frontera OA, Chiari R, Butts C, Wojcik-Tomaszewska J, Coudert B, Garassino MC, Ready N, Felip E, Garcia MA, Waterhouse D, Domine M, Barlesi F, Antonia S, Wohlleber M, Gerber DE, Czyzewicz G, Spigel DR, Crino L, Eberhardt WEE, Li A, Marimuthu S, Brahmer J. Five-Year Outcomes From the Randomized, Phase III Trials CheckMate 017 and 057: Nivolumab Versus Docetaxel in Previously Treated Non-Small-Cell Lung Cancer. J Clin Oncol. 2021 Mar 1;39(7):723-733. doi: 10.1200/JCO.20.01605. Epub 2021 Jan 15. PMID 33449799
- [Background] Armand P, Engert A, Younes A, Fanale M, Santoro A, Zinzani PL, Timmerman JM, Collins GP, Ramchandren R, Cohen JB, De Boer JP, Kuruvilla J, Savage KJ, Trneny M, Shipp MA, Kato K, Sumbul A, Farsaci B, Ansell SM. Nivolumab for Relapsed/Refractory Classic Hodgkin Lymphoma After Failure of Autologous Hematopoietic Cell Transplantation: Extended Follow-Up of the Multicohort Single-Arm Phase II CheckMate 205 Trial. J Clin Oncol. 2018 May 10;36(14):1428-1439. doi: 10.1200/JCO.2017.76.0793. Epub 2018 Mar 27. PMID 29584546
- [Background] Abramson JS, Palomba ML, Gordon LI, Lunning MA, Wang M, Arnason J, Mehta A, Purev E, Maloney DG, Andreadis C, Sehgal A, Solomon SR, Ghosh N, Albertson TM, Garcia J, Kostic A, Mallaney M, Ogasawara K, Newhall K, Kim Y, Li D, Siddiqi T. Lisocabtagene maraleucel for patients with relapsed or refractory large B-cell lymphomas (TRANSCEND NHL 001): a multicentre seamless design study. Lancet. 2020 Sep 19;396(10254):839-852. doi: 10.1016/S0140-6736(20)31366-0. Epub 2020 Sep 1. PMID 32888407